CLINICAL TRIAL: NCT01871389
Title: Impact of Monthly High Dose Oral Cholecalciferol on Serum 25 Hydroxy Vitamin D Levels in Bariatric Surgery Subjects
Status: Completed | Type: Observational
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Lee Mallory Boylan, Professor, Texas Tech University
Other Study IDs: Vitamin D3
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Bariatric Surgery

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- cholecalciferol
- usual treatment

SUMMARY:
Vitamin D deficiency is common after bariatric surgery. This study is designed to determine if a high dose monthly supplement of vitamin D 3 will be effective in helping improve vitamin D status after surgery such as gastric bypass. Bariatric surgery subjects taking monthly high dose cholecalciferol supplements in addition to the standard vitamin D protocol will have a significant rise in serum vitamin D levels compared to the subjects taking only the usual vitamin D protocol.

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese meeting criteria for gastric bypass over age 18

Exclusion Criteria:

* taking medications that affect vitamin D status, elevated serum hydroxy vit D or calcium

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2012-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Serum 25(OH)D3 | Change at 3 and 6 mos

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Bariatric Surgery Center, Lubbock, Texas, United States